CLINICAL TRIAL: NCT05587387
Title: Change of Treatment Landscape and Survival in Metastatic Pancreatic Cancer After Nal-IRI in Republic of Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0776
Record Dates: First submitted 2022-09-26; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Without Nal-IRI/FL; From Jan. 2012 to Jan. 2018 (Before launch of nal-IRI)
- Cohort 2: With Nal-IRI/FL; From Jan. 2018 to Dec. 2021 (After launch of nal-IRI)

SUMMARY:
Pancreatic cancer is a very aggressive disease and its prognosis is poor. Large proportion of patients diagnosed with pancreatic cancer is already in metastatic or locally advanced phases. Although there have been huge improvements in survival for many other cancers over the last few decades, the same isn't true for pancreatic cancer. Median 5-year survival rate for pancreatic cancer is around 10% and there are limited number of treatments approved for pancreatic cancer.

There is no definite consensus on the best second-line chemotherapy for patients with metastatic pancreatic cancer who have progressed after first-line chemotherapy. The randomized phase III study, NAPOLI-1 trial has revealed that liposomal irinotecan (nal-IRI) plus fluorouracil/leucovorin (FL) regimen could be an acceptable treatment option in patients with metastatic pancreatic cancer who had been previously treated with gemcitabine-based chemotherapy.

In this study, The investigators will evaluate how the treatment landscape has been changed since the appearance of nal-IRI in Korea. By retrospectively comparing treatment efficacy and safety outcomes before (cohort 1; without nal-IRI/FL) and after the launch of nal-IRI (cohort 2; with nal-IRI/FL), investigators will identify the degree of improvement in treatment outcome brought about by nal-IRI and will confirm whether the nal-IRI could be applied as an effective treatment option in patients with metastatic pancreatic cancer who failed first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients initially diagnosed as locally advanced pancreatic cancer or metastatic pancreatic cancer and received chemotherapy between 2012 and 2021
2. Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas
3. Documented metastatic disease; disease status may be measurable or non-measurable as defined by RECIST v1.1 guidelines
4. Locally advanced pancreatic cancer; disease status was defined by NCCN guidelines.
5. Recovered from the effects of any prior surgery, radiotherapy, or other antineoplastic therapy
6. At least 18 years of age

Exclusion Criteria:

1. Other histology (ex. Neuroendocrine tumor, etc.)
2. Cohort 2 (other regimens); Patients who received nal-IRI at least once after diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In multiple medicatl center, such as Sinchon Severance hospital, Gangnam Severance hospital, Gachon University Gil hospital and Konkuk University hospital, investigators will collect the medical information according to inclusion criteria and exclusion criteria from 2012 to 2021.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-27 (Estimated); Study Completion 2023-07-27 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS1) | The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. (Up to 100 weeks)
  the duration from diagnosis of pancreatic cancer to death or last follow-up
  - OS1 : the duration from diagnosis of pancreatic cancer to death or last follow-up
Overall survival (OS 2) | The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive. (Up to 100 weeks)
  the duration from nal-IRI treatment initiation to death or last follow-up

SECONDARY OUTCOMES:
Progression free survival | The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse (Up to 100 weeks)
  the duration from treatment initiation to disease progression
Objective response rate | The assessment of the tumor burden after a given treatment in patients with solid tumors and has a long history(Up to 100 weeks)
  the ratio of complete remission and partial remission
Disease control rate | the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.(Up to 100 weeks)
  the ratio of complete remission, partial remission and stable disease
Adverse event | Any undesirable experience associated with the use of a medical product in a patient.(Up to 100 weeks)
  adverse event during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seungmin Bang, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No